CLINICAL TRIAL: NCT04085159
Title: Immunotherapy Targeting Neurofibromatosis or Schwannomatosis
Brief Title: Immunotherapy Based on Antigen-specific Immune Effector Cells Targeting Neurofibromatosis or Schwannomatosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other); Shenzhen Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-19006
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Cancer
Keywords: immunotherapy T cell cancer gene therapy
MeSH Terms: conditions — Neoplasms | interventions — S-1,2-dichlorovinyl-N-acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART/CTL/DCvac cells to treat cancer (Experimental)
  Interventions: Biological: Antigen-specific T cells CART/CTL and DCvac

INTERVENTIONS:
Biological: Antigen-specific T cells CART/CTL and DCvac — Antigen-specific T cells CART/CTL and DCvac cells to treat cancer

SUMMARY:
The primary objective of this study is to verify the safety of antigen-specific T cells (CAR-T) and engineered immune effector cytotoxic T cells (EIE) modified by immunoregulatory genes and immune modified dendritic cell vaccine (DCvac) in the treatment of neurofibromatosis or schwannoma.

DETAILED DESCRIPTION:
Neurofibromatosis (NF) is caused by a genetic change that tends to develop benign tumors around nerves. NF is a lifelong condition that affects all populations equally, regardless of gender or ethnicity. Neurofibromatosis has been classified into three distinct types: NF1, NF2, and schwannomatosis. The hallmark tumors seen in NF2 are vestibular schwannomas, formerly known as acoustic neuromas. Vestibular schwannomas are benign tumors made up of abnormal Schwann cells, which are the cells that give the nerves the lining and insulation needed to conduct information. Vestibular schwannomas can cause hearing loss in one or both ears, depending on whether the tumors are unilateral or bilateral.

Schwannomatosis is the same type of tumor as that of NF2 patients. Tumors are all related to Schwann cells. There is no cure for NF or schwannomatosis. Surgery is the only clinical method at present, and no drugs have been proved to be effective in the treatment of these tumors.

Adoptive immunotherapy based on cytotoxic T lymphocytes reactive with specific antigens has proven to be effective. In vitro induction of tumor antigen-specific immune cells and engineering of target specific immune cells have great potential for cancer eradication. If CAR-T/CTL immunotherapy is effective, it is expected that Neurofibromatosis or Schwannomatosis tumors should shrink or disappear completely. However, the minimal residual tumor cells or cancer stem cells may exist and cause relapse to other tissues and organs. Follow-up immunotherapy must focus on enhancing the anti-tumor immunity. Therefore, this protocol includes follow-up application of DCvac to prevent recurrence. This study proposes a novel protocol of immunotherapy to evaluate the safety and effectiveness of targeting tumor antigens in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent obtained prior to any study-specific procedures.
2. Diagnosis of neurofibromatosis, or schwannomatosis
3. The results of immune staining of the patient's cancer specimens positive for any one or more of a list of tumor-associated antigens.
4. Age ≥ 1 years
5. At least one volumetrically measurable and ≥ 0.5 cc NF-related tumor (schwannoma, ependymoma, meningioma - histological confirmation not required) with radiographic evidence of progression (either as unequivocal progression on conventional MRI, or a >10% volume increase by 3D volumetrics) over the past ≤12 months, designated as the primary target tumor OR Volumetrically measurable and ≥ 0.5 cc VS with ipsilateral progressive hearing loss over the past ≤12 months, designated as the primary target tumor.
6. Progressive Hearing Loss Criteria for Enrollment: Audiogram showing drop in pure tone average (PTA) of 10dB HL at ≥ 2 nonconsecutive or consecutive frequencies or drop in speech discrimination score (SDS) below the 95% critical difference threshold, compared to previous audiogram ≤ 1 year prior.
7. Karnofsky/Lansky performance status (PS) 50-100%. Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
8. Any neurologic deficits must be stable for ≥ 1 week.
9. Adequate bone marrow reserve with

   * absolute neutrophil count (ANC) ≥ 1000/mm3.
   * Platelets ≥100,000/mm3.
10. Adequate renal and hepatic function with

    * Serum creatinine ≤ 2 x upper limit of normal (ULN).
    * Serum bilirubin ≤ 2 x ULN.
    * aspartate aminotransferase (AST)/ALT ≤ 2 x ULN.
    * Alkaline phosphatase ≤ 5 x ULN.
    * Serum bilirubin 2.0 is acceptable in the setting of known Gilbert's syndrome.

Exclusion Criteria:

1. The results of immune staining of the patient's tumor-associated antigens are all negative.
2. Participation in any other cell therapy protocols within one year.
3. Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug.
4. Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study.
5. Pregnant or lactating females.
6. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
7. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

   * Symptomatic congestive heart failure of New York heart Association Class III or IV
   * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
   * severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
   * uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN (Note: Optimal glycemic control should be achieved before starting trial therapy.)
   * active (acute or chronic) or uncontrolled severe infections
   * liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
8. Inadequate bone marrow function:

   * Absolute neutrophil count < 1.0 x 10e9/L.• Platelet count < 100 x 10e9/L.
   * Hb < 9 g/dL.
9. Inadequate liver and renal function:

   * Serum (total) bilirubin > 1.5 x ULN.
   * AST & ALT > 2.5 x ULN (> 5 x ULN in patients with liver metastases).
   * Alkaline phosphatase > 2.5 x ULN (or > 5 x ULN in case of liver metastases or > 10 x ULN in case of bone metastases).
   * Serum creatinine >2.0 mg/dl (> 177 μmol/L).
   * Urine dipstick for protein uria should be < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < 1 g of protein/24 hr.
10. Subject infected with HIV (HIV antibody positive), Treponema pallidum antibody positive or TB culture positive.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse effects after CART/CTL/DCvac cells injection | up to one month
  To assess the safety of autologous CART/CTL/DCvac cells in patients. The percentage of patients who have adverse effects will be evaluated by using the NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Rate of successful CART/CTL/DCvac cell production | up to one month
  The percentage of successful CART/CTL/DCvac cell generation, which is based on products which pass the safety test after standard culture procedures, viable for at least one preparation, will be evaluated.
Ability of CART/CTL/DCvac cells to induce anti-cancer reaction | after 1 month from CART/CTL/DCvac cells infusion until 12 months after infusion
  measurement of concentration of tumor associated markers
Ability of CART/CTL/DCvac cells for anti-tumor reaction | after 1 month from CART/CTL/DCvac cells infusion until 24 months after infusion
  Objective response (complete response (CR) + partial response (PR)) was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Department of Neurosurgery, Shenzhen Hospital, Southern Medical University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No